CLINICAL TRIAL: NCT02927132
Title: Guilt and Expressive Writing for Reducing Alcohol Use in College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Clayton Neighbors, Professor, Director of the Social Influences and Health Behaviors Lab, University of Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 3660702; 1R01AA023495-01 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-10-06 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Alcohol Consumption
Keywords: Drinking, Alcohol
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- Alcohol-Guilt Condition (Experimental): In this condition, participants are asked to write about an incident in which they drank heavily and experienced guilt.
  Participants in this condition will come into the lab one time each week for three weeks to complete the writing task. They will then complete follow-up surveys remotely, at 1 month, 3 months, 6 months, and 12 months.
  Interventions: Behavioral: Expressive Writing
- Distress-Guilt Condition (Experimental): In this condition, participants are asked to write about an upsetting incident where they experienced guilt.
  Participants in this condition will come into the lab one time each week for three weeks to complete the writing task. They will then complete follow-up surveys remotely, at 1 month, 3 months, 6 months, and 12 months.
  Interventions: Behavioral: Expressive Writing
- Alcohol-No Guilt Condition (Experimental): In this condition, participants are asked to write about a negative drinking incident that they had experienced.
  Participants in this condition will come into the lab one time each week for three weeks to complete the writing task. They will then complete follow-up surveys remotely, at 1 month, 3 months, 6 months, and 12 months.
  Interventions: Behavioral: Expressive Writing
- Distress-No Guilt Condition (Experimental): In this condition, participants are asked to write about an upsetting experience that has affected their life.
  Participants in this condition will come into the lab one time each week for three weeks to complete the writing task. They will then complete follow-up surveys remotely, at 1 month, 3 months, 6 months, and 12 months.
  Interventions: Behavioral: Expressive Writing
- Neutral Control Condition (No Intervention): In this condition, participants are asked to write about the laboratory room in which they are seated.
  Participants in this condition will come into the lab one time each week for three weeks to complete the writing task. They will then complete follow-up surveys remotely, at 1 month, 3 months, 6 months, and 12 months.
- Personalized Normative Feedback (Experimental): Participants in the PNF condition will be given gender-specific personalized feedback regarding their alcohol use. Participants will be presented with the drinking estimates that they previously gave in addition to average gender-specific drinking estimates provided by 1124 students at the University of Houston. Feedback will be provided for drinking frequency (i.e., number of drinking days per week), and drinking quantity (i.e., the number of drinks consumed per week and number of drinks consumed per typical drinking occasion). Participants will also receive a printed a copy of the feedback for their records. PNF participants will receive feedback immediately after the baseline assessment. We also wanted to control for any differences that might be attributed to attention. Thus, participants will be scheduled to come in to the lab for two more sessions, during which time they will write about the laboratory room in which they are seated.
  Interventions: Behavioral: Personalized Normative Feedback

INTERVENTIONS:
Behavioral: Expressive Writing — Expressive writing is a brief intervention that has been linked to various health and social benefits. Expressing emotions through writing can lead to decreased levels of stress and negative affect, thereby serving as a coping mechanism. Furthermore, expressive writing allows participants to reconstruct their traumatic experiences and reorganize their memory of these events into a narrative. Expressive writing has been used to target drinking. Research has found that students have reduced drinking intentions after writing about a negative drinking event compared to control,suggesting that a narrative intervention may be effective in reducing drinking. Other research suggests that feelings of guilt were more strongly associated with intentions to reduce drinking after writing about a negative drinking event, and that this event-related guilt mediated intervention effects.
  Arms: Alcohol-Guilt Condition; Alcohol-No Guilt Condition; Distress-Guilt Condition; Distress-No Guilt Condition
Behavioral: Personalized Normative Feedback — PNF approaches use information designed to correct normative misperceptions to reduce heavy drinking. Three pieces of information are necessary when providing personalized normative feedback: information about a student's own drinking, information about the student's perceptions of others' drinking, and information about others' actual drinking. The presentation of this information is designed to change students' perceptions of "normal" drinking by exposing their misperceptions of the norm as well as by comparing their behavior with "normal" behavior.
  Arms: Personalized Normative Feedback

SUMMARY:
This research seeks to evaluate expressive writing as a novel intervention for problem drinking among college students. The vast majority of individually focused brief interventions targeting college drinking have focused on personalized feedback approaches and recent innovations have largely been limited to finer distinctions of these, which require assessment and programming for implementation. The present research proposes expressive writing as a novel alternative, which has been used extensively in other domains but not as an alcohol intervention strategy.

H1a: Participants writing about negative drinking events will show reduced drinking and drinking-related negative consequences relative to students in the neutral control group.

H1b: Participants writing about distressing non-alcohol events will show increased psychological wellbeing relative to students in the neutral control group.

H1c: Participants writing about negative drinking events will show reduced drinking and consequences compared with an empirically-supported brief intervention (i.e., PNF). This is an exploratory hypothesis.

H2a: Alcohol narratives will have stronger effects on alcohol outcomes relative to distress narratives.

H2b: Alcohol guilt narratives will have the strongest effect on alcohol outcomes relative to all other conditions.

H3a: Expression of guilt, assessed by self-report and by content coding with LIWC, will mediate intervention effects on drinking outcomes.

H3b: Change thought, assessed by LIWC coding, will mediate intervention effects on drinking.

DETAILED DESCRIPTION:
The current research builds on previous research targeting heavy drinking among college students. A large volume of research has provided an impressive data base supporting one type of individually-focused alcohol intervention for this population (i.e., personalized feedback). The success of this paradigm has probably contributed to the dearth of consideration of alternative paradigms. Expressive writing is one such alternative, which has received extensive support in other domains but has only recently been considered as a potential intervention for heavy drinking. The preliminary data examining this approach is promising and provides a firm foundation for this efficacy trial. Further, this research incorporates novel theoretical constructs including the specific focus on guilt in expressive writing content as well as "change thought," as an analogue to the mechanism presumed to underlie motivational treatments for alcohol and other substance use disorders. The investigators plan to employ similar methods which have been used successfully in other large NIAAA funded trials evaluating brief interventions for heavy drinking college students.

This research consists of an intervention study to evaluate expressive writing as a brief intervention in reducing drinking and improving psychological well-being among college students. Participation in the study involves completion of a screening assessment, a baseline assessment, the intervention procedure, post-intervention assessment, and follow-up assessments at 1-, 3-, 6-, and 12-months. Heavy drinking college students (N = 600) will be randomly assigned to one of six conditions based on the 2 (alcohol vs. distress topics) × 2 (guilt vs. no guilt focus) + 1 (neutral control) + 1 (personalized normative feedback) design. Before completing the baseline survey, students will be randomly assigned to one of six study conditions, five of which involve writing during three sessions over the course of one month. Specifically, participants will be assigned to write about a heavy drinking event, a heavy drinking event that elicited guilt, a distressing event, a distressing event that elicited guilt, or their first day of college (neutral control condition).

Participants randomly assigned to the PNF condition will receive traditional personalized normative feedback regarding how their drinking compares with other students of the same gender at the university. The norms will come from a large recently completed alcohol survey conducted at the University of Houston examining social norms and alcohol prevention (R01AA014576). To maintain consistency across conditions, participants in the PNF condition will still come into the lab three times. They will receive feedback during the first intervention session and will be asked to complete the same narrative prompts as the neutral control condition for their second and third session. For individuals in the expressive writing conditions, there will be three narrative prompts to complete every week for three weeks, the first of which will occur following the baseline assessment. All baseline assessments, narrative intervention assignments, and immediate post-tests for all conditions will be conducted in-lab. All other assessments including screening and follow-up assessments will be completed remotely by web. The rationale for including a personalized normative feedback condition is to be able to compare the efficacy of expressive writing interventions with existing brief alcohol interventions. Thus, the present design allows not only for evaluation of efficacy relative to a control condition but also will evaluate comparative efficacy relative to an existing empirically-supported brief alcohol intervention.

Aims will be evaluated using multi-level regression analyses, often referred to as Hierarchical Linear Modeling (HLM) or mixed-effects modeling. With respect to evaluating main effects of experimental conditions on drinking, each participant will provide baseline, post-intervention, 1-month, 3-month, 6-month, and 12-month follow-up data. Hypotheses will be tested using specific contrast vectors, using a general linear hypothesis framework. The study consists of a (2×2+1+1) design, represented as a factorial design with the addition of a control group that will write about their first day of school and a computer-based PNF comparison group. Hypotheses will be tested with contrasts corresponding to the questions of interest. The first two hypotheses represent contrasts between the alcohol narrative conditions and the neutral control condition (H1a) and between the guilt narrative conditions and the neutral control condition (H1b). In examining these hypotheses, the investigators will construct two dummy coded variables reflecting alcohol versus non-alcohol narratives conditions and between guilt and non-guilt narrative conditions with the reference group being the neutral control condition. Thus, the PNF group will not be included in the tests of these two hypotheses. Dependent variables will include alcohol outcomes for H1a and psychological well-being for H1b. For these analyses each participant will provide up to 5 repeated measures (i.e., baseline, 1-month, 3-months, 6-months, and 12-months), yielding up to 3000 Level 1 cases (repeated-measures) across 600 Level 2 cases.

The investigators will also evaluate mediators of intervention effects. Additionally, the investigators will follow procedures to assess mediation. Mediation will test indirect effects using the AB products method where A will represent effects of intervention contrasts by time interactions on mediators (expression of guilt and change thought). B will represent the associations of mediators on subsequent drinking outcomes. Both A and B paths will control for baseline outcomes. Evaluation of hypotheses regarding the moderation effect will test whether individual differences in guilt-proneness interact with intervention contrasts. These will be tested by expanding the above model to add main effects and product terms of proposed moderators with intervention contrasts.

Power analyses focus on estimating a sample size large enough to detect "true" effects, thereby avoiding Type II errors. Sample size estimates were obtained for intervention contrasts. Necessary sample sizes were assessed via sample size and power equations for normally distributed outcomes. Effect-sizes and variance components were based on preliminary studies, and power was set at 0.80 for all estimates. Power was estimated using the Optimal Design software program. The investigators anticipate intervention effects relative to the neutral control condition on drinking to be in the range of delta =.30-.40). Based on the proposed sample size of 500 (~PNF not included in H1a and H1b), given five assessment points, the investigators anticipate the ability to detect main effects of intervention contrasts with power=.80. Considering maximum anticipated attrition rates of 20% the investigators will have .80 power to detect effects sizes of delta = .28 and greater.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the screening survey include

* Being between 18-26 years of age
* Being a registered UH student.

Inclusion criteria for longitudinal participation include

* Scoring 5+ and 7+ on the AUDIT-C for women/men respectively
* Being 18-26 years of age
* Being a registered UH student
* Providing consent to participate in the study

Exclusion Criteria:

Exclusion criteria for the screening survey include

* Not meeting inclusion criteria (i.e., not between 18-26 years of age, not a registered UH student)or unwillingness to participate.

Exclusion criteria for baseline include

* Not meeting any of the inclusion criteria, unwillingness to participate, and failure to provide consent.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Consumption measured by The Timeline Follow-Back (TLFB) | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  The TLFB is a calendar based measure assessing daily drinking (and abstinence) over a designated period of time.
  Number of drinks in the past month will be calculated as the sum of drinks recorded each day of the past month on the TLFB.
Change in Drinking Intentions as measured by a modified version of the Daily Drinking Questionnaire (DDQ). | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  Response options will be identical to the DDQ, but participants will be asked to indicate their intended drinking behaviors.
  Participants fill in the average number of standard drinks they intend to consume for each day of the week over the next month. Typical number of intended drinks per week will be calculated as the sum of typical number of drinks intended per day on the Daily Drinking Questionnaire.
Change in Alcohol Consumption measured by Alcohol Use Disorders Identification Test (AUDIT). | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  The AUDIT assesses for hazardous alcohol use, dependence symptoms, and harmful use. Scores for each question range from 0 to 4, with the first response for each question (e.g. never) scoring 0, the second (e.g. less than monthly) scoring 1, the third (e.g. monthly) scoring 2, the fourth (e.g. weekly) scoring 3, and the last response (e.g. daily or almost daily) scoring 4. For questions 9 and 10, which only have three responses, the scoring is 0, 2 and 4 (from left to right). A score of 8 or more is associated with harmful or hazardous drinking.
Change in Alcohol Consumption measured by Quantity-Frequency-Peak Alcohol Use Index. | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  The Quantity-Frequency-Peak Alcohol Use Index is a five-item questionnaire that includes two items addressing the occasion where respondents drank the most during the previous three months, two items addressing typical weekend drinking in the previous three months, and one item addressing typical number of drinking days per week in the previous three months. Drinking frequency will be assessed by item #5 of the Quantity/Frequency Questionnaire, which asks how many days during the past week participants have consumed alcohol.
Change in Alcohol Consumption measured by the Daily Drinking Questionnaire (DDQ. | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  Typical weekly drinking and typical drinks per occasion will be assessed with the DDQ. Participants fill in the average number of standard drinks they consumed and the time period of consumption for each day of the week over the previous three months. Typical number of drinks per week will be calculated as the sum of typical number of drinks per day on the Daily Drinking Questionnaire.
Change in Drinking Intentions as measured by a modified version of the Quantity-Frequency-Peak Alcohol Use Index (QF). | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  Response options will be identical to the QF, but participants will be asked to indicate their intended drinking behaviors. Intended drinking frequency will be assessed by item #5 of the Quantity/Frequency Questionnaire, which asks how many days during the next week participants intend to consume alcohol.
Changes in Psychological Well-being Outcomes as measured by the Center for Epidemiological Studies Depression Scale (CES-D) | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  Depression will be assessed by the Ces-D, a 20-item measure of depressive symptomatology in the general population. Answers are on a scale of 1 (rarely) to 4 (most or all of the time). A score of 11 is indicative of significant or mild depressive symptomology, and higher scores are indicative of greater symptoms.
Changes in Psychological Well-being Outcomes as measured by Positive and Negative Affect Scale (PANAS) | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  Mood will be assessed by the PANAS, a 22-item measure of the degree to which one experiences positive and negative affective states on a regular basis.
  For a positive affect score, items 1 (interested), 3 (excited), 5 (strong), 9 (enthusiastic), 10 (proud), 12 (alert), 14 (inspired), 16 (determined), 17 (attentive), and 19 (active) will be added, with higher scores representing higher levels of positive affect.
  For a negative affect score, items 2 (distressed), 4 (upset), 6 (guilty), 7 (scared), 8 (hostile), 11 (irritable), 13 (ashamed), 15 (nervous), 18 (jittery) and 20 (afraid) will be added, with lower scores representing lower levels of negative affect.
Changes in Psychological Well-being Outcomes as measured by Satisfaction with Life Scale (SWLS). | Baseline, 1 month follow-up, 3 month follow-up, 6 month follow-up, 12 month follow-up
  This short, 5-item measure is designed to measure cognitive judgments of satisfaction with one's life. Each item is rated on a scale of 1 (strongly disagree) to 7 (strongly agree). A score of 31-35 indicates that a participant is extremely satisfied, a score of 26-30 indicates that a participant is satisfied, a score of 21-25 indicates that a participant is slightly satisfied, a score of 20 indicates that a participant is neutral, a score of 15-19 indicates that a participant is slightly dissatisfied, a score of 10-14 indicates that a participant is dissatisfied, and a score of 5-9 indicates that a participant is extremely dissatisfied.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ames SC, Patten CA, Offord KP, Pennebaker JW, Croghan IT, Tri DM, Stevens SR, Hurt RD. Expressive writing intervention for young adult cigarette smokers. J Clin Psychol. 2005 Dec;61(12):1555-70. doi: 10.1002/jclp.20208. PMID 16193479
- [Background] Ames SC, Patten CA, Werch CE, Schroeder DR, Stevens SR, Fredrickson PA, Echols JD, Pennebaker JW, Hurt RD. Expressive writing as a smoking cessation treatment adjunct for young adult smokers. Nicotine Tob Res. 2007 Feb;9(2):185-94. doi: 10.1080/14622200601078525. PMID 17365749
- [Background] Amrhein PC, Miller WR, Yahne CE, Palmer M, Fulcher L. Client commitment language during motivational interviewing predicts drug use outcomes. J Consult Clin Psychol. 2003 Oct;71(5):862-78. doi: 10.1037/0022-006X.71.5.862. PMID 14516235
- [Background] Baer JS, Marlatt GA, Kivlahan DR, Fromme K, Larimer ME, Williams E. An experimental test of three methods of alcohol risk reduction with young adults. J Consult Clin Psychol. 1992 Dec;60(6):974-9. doi: 10.1037//0022-006x.60.6.974. PMID 1460160
- [Background] Baikie KA, Geerligs L, Wilhelm K. Expressive writing and positive writing for participants with mood disorders: an online randomized controlled trial. J Affect Disord. 2012 Feb;136(3):310-9. doi: 10.1016/j.jad.2011.11.032. Epub 2011 Dec 30. PMID 22209127
- [Background] Barclay LJ, Skarlicki DP. Healing the wounds of organizational injustice: examining the benefits of expressive writing. J Appl Psychol. 2009 Mar;94(2):511-23. doi: 10.1037/a0013451. PMID 19271805
- [Background] Barnett NP, Goldstein AL, Murphy JG, Colby SM, Monti PM. "I'll never drink like that again": characteristics of alcohol-related incidents and predictors of motivation to change in college students. J Stud Alcohol. 2006 Sep;67(5):754-63. doi: 10.15288/jsa.2006.67.754. PMID 16847545
- [Background] Carey KB, Scott-Sheldon LA, Carey MP, DeMartini KS. Individual-level interventions to reduce college student drinking: a meta-analytic review. Addict Behav. 2007 Nov;32(11):2469-94. doi: 10.1016/j.addbeh.2007.05.004. Epub 2007 May 17. PMID 17590277
- [Background] Carey KB, Scott-Sheldon LA, Elliott JC, Bolles JR, Carey MP. Computer-delivered interventions to reduce college student drinking: a meta-analysis. Addiction. 2009 Nov;104(11):1807-19. doi: 10.1111/j.1360-0443.2009.02691.x. Epub 2009 Sep 10. PMID 19744139
- [Background] Chung CK, Pennebaker JW. Variations in the spacing of expressive writing sessions. Br J Health Psychol. 2008 Feb;13(Pt 1):15-21. doi: 10.1348/135910707X251171. PMID 18230224
- [Background] Collins SE, Carey KB. The theory of planned behavior as a model of heavy episodic drinking among college students. Psychol Addict Behav. 2007 Dec;21(4):498-507. doi: 10.1037/0893-164X.21.4.498. PMID 18072832
- [Background] Collins SE, Carey KB, Sliwinski MJ. Mailed personalized normative feedback as a brief intervention for at-risk college drinkers. J Stud Alcohol. 2002 Sep;63(5):559-67. doi: 10.15288/jsa.2002.63.559. PMID 12380852
- [Background] Craft MA, Davis GC, Paulson RM. Expressive writing in early breast cancer survivors. J Adv Nurs. 2013 Feb;69(2):305-15. doi: 10.1111/j.1365-2648.2012.06008.x. Epub 2012 Apr 11. PMID 22494086
- [Background] Cronce, J. M., & Larimer, M. E. (2012). Brief individual-focused alcohol interventions for college students. In H. White, D. L. Rabiner (Eds.), College drinking and drug use (pp. 161-183). New York, NY US: Guilford Press.
- [Background] Dearing RL, Stuewig J, Tangney JP. On the importance of distinguishing shame from guilt: relations to problematic alcohol and drug use. Addict Behav. 2005 Aug;30(7):1392-404. doi: 10.1016/j.addbeh.2005.02.002. Epub 2005 Apr 13. PMID 16022935
- [Background] Doumas, D. M., Kane, C. M., Navarro, B. B., & Roman, J. (2011). Decreasing heavy drinking in first-year students: Evaluation of a web-based personalized feedback program administered during orientation. Journal of College Counseling, 14(1), 5-20. doi:10.1002/j.2161-1882.2011.tb00060.x
- [Background] Elliott JC, Carey KB, Bolles JR. Computer-based interventions for college drinking: a qualitative review. Addict Behav. 2008 Aug;33(8):994-1005. doi: 10.1016/j.addbeh.2008.03.006. Epub 2008 Apr 7. PMID 18538484
- [Background] Francis ME, Pennebaker JW. Putting stress into words: the impact of writing on physiological, absentee, and self-reported emotional well-being measures. Am J Health Promot. 1992 Mar-Apr;6(4):280-7. doi: 10.4278/0890-1171-6.4.280. PMID 10146806
- [Background] Gaume J, Bertholet N, Faouzi M, Gmel G, Daeppen JB. Does change talk during brief motivational interventions with young men predict change in alcohol use? J Subst Abuse Treat. 2013 Feb;44(2):177-85. doi: 10.1016/j.jsat.2012.04.005. Epub 2012 Jun 1. PMID 22658289
- [Background] Harvey AG, Farrell C. The efficacy of a Pennebaker-like writing intervention for poor sleepers. Behav Sleep Med. 2003;1(2):115-24. doi: 10.1207/S15402010BSM0102_4. PMID 15600133
- [Background] Klein K, Boals A. Expressive writing can increase working memory capacity. J Exp Psychol Gen. 2001 Sep;130(3):520-33. doi: 10.1037//0096-3445.130.3.520. PMID 11561925
- [Background] Larimer ME, Cronce JM. Identification, prevention, and treatment revisited: individual-focused college drinking prevention strategies 1999-2006. Addict Behav. 2007 Nov;32(11):2439-68. doi: 10.1016/j.addbeh.2007.05.006. Epub 2007 May 17. PMID 17604915
- [Background] Larimer ME, Lee CM, Kilmer JR, Fabiano PM, Stark CB, Geisner IM, Mallett KA, Lostutter TW, Cronce JM, Feeney M, Neighbors C. Personalized mailed feedback for college drinking prevention: a randomized clinical trial. J Consult Clin Psychol. 2007 Apr;75(2):285-93. doi: 10.1037/0022-006X.75.2.285. PMID 17469886
- [Background] Labrie JW, Lewis MA, Atkins DC, Neighbors C, Zheng C, Kenney SR, Napper LE, Walter T, Kilmer JR, Hummer JF, Grossbard J, Ghaidarov TM, Desai S, Lee CM, Larimer ME. RCT of web-based personalized normative feedback for college drinking prevention: are typical student norms good enough? J Consult Clin Psychol. 2013 Dec;81(6):1074-86. doi: 10.1037/a0034087. Epub 2013 Aug 12. PMID 23937346
- [Background] Leith, K. P., & Baumeister, R. F. (1998). Empathy, shame, guilt, and narratives of interpersonal conflicts: Guiltprone people are better at perspective taking. Journal of Personality, 66, 1-37.
- [Background] Lewis MA, Neighbors C. Optimizing personalized normative feedback: the use of gender-specific referents. J Stud Alcohol Drugs. 2007 Mar;68(2):228-37. doi: 10.15288/jsad.2007.68.228. PMID 17286341
- [Background] Lewis MA, Neighbors C, Oster-Aaland L, Kirkeby BS, Larimer ME. Indicated prevention for incoming freshmen: personalized normative feedback and high-risk drinking. Addict Behav. 2007 Nov;32(11):2495-508. doi: 10.1016/j.addbeh.2007.06.019. Epub 2007 Jun 28. PMID 17658695
- [Background] Lu Q, Stanton AL. How benefits of expressive writing vary as a function of writing instructions, ethnicity and ambivalence over emotional expression. Psychol Health. 2010 Jul;25(6):669-84. doi: 10.1080/08870440902883196. PMID 20204944
- [Background] Lumley, M. A., & Provenzano, K. M. (2003). Stress management through written emotional disclosure improves academic performance among college students with physical symptoms. Journal of Educational Psychology, 95(3), 641-649. doi:10.1037/0022 0663.95.3.641
- [Background] Miller MB, Leffingwell T, Claborn K, Meier E, Walters S, Neighbors C. Personalized feedback interventions for college alcohol misuse: an update of Walters & Neighbors (2005). Psychol Addict Behav. 2013 Dec;27(4):909-20. doi: 10.1037/a0031174. Epub 2012 Dec 31. PMID 23276309
- [Background] Neighbors C, Larimer ME, Lewis MA. Targeting misperceptions of descriptive drinking norms: efficacy of a computer-delivered personalized normative feedback intervention. J Consult Clin Psychol. 2004 Jun;72(3):434-47. doi: 10.1037/0022-006X.72.3.434. PMID 15279527
- [Background] Neighbors C, Lewis MA, Bergstrom RL, Larimer ME. Being controlled by normative influences: self-determination as a moderator of a normative feedback alcohol intervention. Health Psychol. 2006 Sep;25(5):571-9. doi: 10.1037/0278-6133.25.5.571. PMID 17014274
- [Background] Neighbors C, Lee CM, Lewis MA, Fossos N, Walter T. Internet-based personalized feedback to reduce 21st-birthday drinking: a randomized controlled trial of an event-specific prevention intervention. J Consult Clin Psychol. 2009 Feb;77(1):51-63. doi: 10.1037/a0014386. PMID 19170453
- [Background] Neighbors C, Lewis MA, Atkins DC, Jensen MM, Walter T, Fossos N, Lee CM, Larimer ME. Efficacy of web-based personalized normative feedback: a two-year randomized controlled trial. J Consult Clin Psychol. 2010 Dec;78(6):898-911. doi: 10.1037/a0020766. PMID 20873892
- [Background] Pennebaker, J. W. (1997). Writing about emotional experiences as a therapeutic process. Psychological Science, 8(3), 162-166. doi:10.1111/j.1467-9280.1997.tb00403.x
- [Background] Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. J Abnorm Psychol. 1986 Aug;95(3):274-81. doi: 10.1037//0021-843x.95.3.274. No abstract available. PMID 3745650
- [Background] Rodriguez LM, Young CM, Neighbors C, Campbell MT, Lu Q. Evaluating guilt and shame in an expressive writing alcohol intervention. Alcohol. 2015 Aug;49(5):491-8. doi: 10.1016/j.alcohol.2015.05.001. Epub 2015 May 18. PMID 26074424
- [Background] Smyth J, Helm R. Focused expressive writing as self-help for stress and trauma. J Clin Psychol. 2003 Feb;59(2):227-35. doi: 10.1002/jclp.10144. PMID 12552631
- [Background] Spera, S. P., Buhrfeind, E. D., & Pennebaker, J. W. (1994). Expressive writing and coping with job loss. Academy of Management Journal, 37(3), 722-733. doi:10.2307/256708
- [Background] Stanton AL, Danoff-Burg S, Sworowski LA, Collins CA, Branstetter AD, Rodriguez-Hanley A, Kirk SB, Austenfeld JL. Randomized, controlled trial of written emotional expression and benefit finding in breast cancer patients. J Clin Oncol. 2002 Oct 15;20(20):4160-8. doi: 10.1200/JCO.2002.08.521. PMID 12377959
- [Background] Walters ST, Neighbors C. Feedback interventions for college alcohol misuse: what, why and for whom? Addict Behav. 2005 Jul;30(6):1168-82. doi: 10.1016/j.addbeh.2004.12.005. Epub 2005 Jan 20. PMID 15925126
- [Background] Young CM, Rodriguez LM, Neighbors C. Expressive writing as a brief intervention for reducing drinking intentions. Addict Behav. 2013 Dec;38(12):2913-7. doi: 10.1016/j.addbeh.2013.08.025. Epub 2013 Sep 4. PMID 24064189
- [Background] Babor, T.F., Higgins-Biddle, J.C., Saunders, J.B., Monteriro, M.G. (2001). AUDIT The alcohol use disordersidentification test: Guidelines for use in primary care. 2nd Edition. WHO/MNH/DAT 89.4, World Health Organization, Geneva.
- [Background] Baer, J. S. (1993). Etiology and secondary prevention of alcohol problems with young adults. In J. Baer, G.Marlatt, R. McMahon (Eds.), Addictive behaviors across the life span: Prevention, treatment, and policy issues (pp. 111-137). Thousand Oaks, CA US: Sage Publications, Inc.
- [Background] Searles JS, Helzer JE, Rose GL, Badger GJ. Concurrent and retrospective reports of alcohol consumption across 30, 90 and 366 days: interactive voice response compared with the timeline follow back. J Stud Alcohol. 2002 May;63(3):352-62. doi: 10.15288/jsa.2002.63.352. PMID 12086136
- [Background] Knee, C., & Neighbors, C. (2002). Self-determination, perception of peer pressure, and drinking among college students. Journal of Applied Social Psychology, 32(3), 522-543.doi:10.1111/j.1559-1816.2002.tb00228.x
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] White HR, Labouvie EW. Towards the assessment of adolescent problem drinking. J Stud Alcohol. 1989 Jan;50(1):30-7. doi: 10.15288/jsa.1989.50.30. PMID 2927120
- [Background] Hurlbut SC, Sher KJ. Assessing alcohol problems in college students. J Am Coll Health. 1992 Sep;41(2):49-58. doi: 10.1080/07448481.1992.10392818. PMID 1460173
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Radloff, L. S. (1977). The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1(3), 385-401.doi:10.1177/014662167700100306
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493